CLINICAL TRIAL: NCT03531580
Title: Brain Images Before and After Upgrade of the MRI-scanner (Siemens Tim TRIO vs Siemens PRISMA FIT) - The TimFit Study
Brief Title: Comparing Brain Images Before and After MRI-upgrade - TimFit Upgrade Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EC/2017/1103
Record Dates: First submitted 2017-11-20; First posted 2018-05-21 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Neuroimaging; Quality Control
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy volunteers (Experimental): six healthy volunteers: 3 male (age 20-40; 40-60 and 60+) and 3 female (age 20-40; 40-60 and 60+)
  Interventions: Device: Magnetic Resonance Imaging

INTERVENTIONS:
Device: Magnetic Resonance Imaging — Brain imaging using magnetic resonance imaging, using several MRI sequences: structural imaging (grey matter, using T1-imaging), cerebral perfusion using arterial spin labeling), functional and effective connectivity (using resting-state functional MRI), white matter tracts (using diffusion imaging), white matter lesions (using Fluid-attenuated inversion recovery MRI (FLAIR)) and microbleeds (using Susceptibility weighted imaging (SWI))

SUMMARY:
In the Ghent University, an upgrade of the MRI-scanner used for research from Siemens Trio Tim to Siemens Prisma Fit is planned in the near future. As a change of MRI hard- and software might influence brain images, it is necessary to evaluate the images before and after the upgrade.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer

Exclusion Criteria:

* Protheses or artificial implants, no magnetic or metal parts in the body
* Being pregnant or breastfeeding
* Having claustrophobia

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in grey matter volume before versus after MRI-upgrade | 7 months, 4 scan sessions of max 1 hour
Change in cerebral perfusion (ml/100g/min) using Arterial Spin Labeling before versus after MRI-upgrade | 7 months, 4 scan sessions of max 1 hour
Change in arterial transit times before versus after MRI-upgrade | 7 months, 4 scan sessions of max 1 hour
Change in functional connectivity (fc) using Resting State functional MRI before versus after MRI-upgrade | 7 months, 4 scan sessions of max 1 hour
Change in effective connectivity using resting state functional MRI before versus after MRI-upgrade | 7 months, 4 scan sessions of max 1 hour
Change in white matter diffusion before versus after MRI-upgrade | 7 months, 4 scan sessions of max 1 hour
Difference in image quality of FLAIR image before versus after MRI-upgrade | 7 months, 4 scan sessions of max 1 hour
Difference in image quality of SWI image before versus after MRI-upgrade | 7 months, 4 scan sessions of max 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Eric Achten, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- Ghent University, Ghent, Belgium